CLINICAL TRIAL: NCT02470052
Title: A Prospective, Open-label, Single-arm, Multicenter Clinical Study to Evaluate the Safety and Effectiveness of the OL-BF-001 for Severe Emphysema
Brief Title: A Prospective Multicenter Clinical Study to Evaluate the Safety and Effectiveness of the OL-BF-001 for Severe Emphysema
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMSC-1401
Record Dates: First submitted 2015-06-05; First posted 2015-06-12 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Emphysema
Keywords: Endobronchial Valves; Intrabronchial Valves; Bronchial Valve; Chronic Obstructive Pulmonary Disease; Pulmonary Disease, Chronic Obstructive; Bronchoscopic Lung Volume Reduction; Emphysema; Pulmonary Emphysema; Lung Diseases; Respiratory Tract Disease
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive; Pulmonary Emphysema; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OL-BF-001 (Experimental): Subjects assigned to this study will undergo a bronchoscopic procedure to have valves placed in the most diseased lobe of the lung to occlude all segments of the lobe. The subjects will also receive medical management.
  Interventions: Device: OL-BF-001

INTERVENTIONS:
Device: OL-BF-001 — Subjects assigned to this study will undergo a bronchoscopic procedure to have valves placed in the most diseased lobe of the lung to occlude all segments of the lobe. The subjects will also receive medical management.

SUMMARY:
This is a multicenter,single-arm,open-label study designed to evaluate improvement of lung function and safety after treatment with OL-BF-001 for severe emphysema.

OL-BF-001 consists of a bronchial valve, deployment catheter, loader and airway sizing kit. A bronchial valve is a small, umbrella-shaped, one-way valve that is placed inside the airways of one lung. It is used to redirect air from the less healthy to the more healthy parts of the lung. This helps to reduce over-inflation and may improve overall lung function and quality of life for people living with emphysema.

ELIGIBILITY:
Inclusion Criteria:

* Subject is treated by maximum medical management（ pharmacological therapy and nonpharmacological therapy ) for 3 months and over before screening testing and the same treatment will be conducted during the study period.
* Subject must have severe dyspnea which is defined as a mMRC ≥ 2.
* Subject's obstructive disease is severe as defined by following post-bronchodilator spirometry values: FEV1/FVC < 70% and 20% of predicted ≤ FEV1 < 50% of predicted
* Subject's hyperinflation is defined by: RV/TLC ≥ 40%
* Subject has severe emphysema and high heterogeneity defined as: a target lobe with ≥ 50% emphysema involvement and clearly different with the ipsilateral lobe, which is judged by visual assessment of thoracic CT. Lung perfusion scan is added to the assessment in principle.
* The target lobe and ipsilateral lobe will be separated with an intact fissure. An intact fissure will be estimated visually to be ≥ 90% complete with no segmental vessels crossing from one lobe to the adjacent lobe.
* Subject must be able to demonstrate physical ability to participate in the study by performing a 6-minute walk distance of ≥ 140 m.
* Subject has abstained from cigarette smoking for 3 months and over before screening testing, and is able to continue to abstain throughout the study.
* Investigator has confirmed that medical management has been conducted enough and disease state has been stable and without a COPD exacerbation for 6 weeks and over before screening testing.
* Subject is able to participate in the study, complete the required follow-up visits, and maintain consistent nutrition and exercise habits during the study period.
* Subject provides informed consent and is willing and able to return for all study examinations.

Exclusion Criteria:

* Subject has a severe gas exchange abnormality in either PaCO2 or PaO2 as defined by: PCO2 > 50 mmHg, or PO2 < 50 mmHg on room air
* Subject with DLCO < 20% of predicted
* Subject has a BMI < 15kg/m2.
* Subject has a risk of thromboembolism.(D-dimer value is used as a reference.)
* Subject had COPD exacerbation which required hospitalization or administration of systemic steroids twice or more in the past 1 year prior to screening testing.
* Subject has a history of pneumothorax twice or more in the past 1 year prior to screening testing.
* Subject has a large amount of sputum production on a daily basis.
* Subject has clinically apparent asthma.
* Subject has giant bulla (> 1/3 volume in either lung. If subject has multiple bullae, the sum of them is judged whether or not > 1/3 volume in either lung. )
* Patient has pulmonary hypertension based upon clinical evaluation.
* Subject uses oral steroids 10 mg/day and over in prednisolone conversion.
* Subject has comorbidities that will limit participation in the study, or follow-up during the study period.
* Subject has a history of thoracic surgeries.
* Subject has thoracic comorbidities (lung nodules, infections(e.g. Pulmonary tuberculosis), Interstitial pneumonia, etc.) , which are anticipated to require evaluation or intervention during the 12 months study period.
* Subject is strongly suspected of pleural adhesions.
* Subject has indicated Left ventricular ejection fraction(LVEF) ≤ 30% within 6 months prior to screening testing. *Subject,who had severe cardiovascular diseases in the past but can control them currently, doesn't meet this criteria.
* Subject is judged as ineligible due to a risk of hemoptysis by investigators.
* Subject has demonstrated unwillingness or inability to complete screening and/or baseline testing.
* Subject has α1-antitrypsin deficiency.
* Subject is classified as ASA Class greater than P4 or has comorbidities that could significantly increase the risk related with bronchoscopy procedure.
* Subject has latex allergy.
* Subject has metallic allergy.
* Subject participated in a study of an investigational drug or device within the 30 days prior to participation in this study, or is currently participating in another clinical study.
* Following women subjects are ineligible: Pregnant women, lactating women, potentially pregnant women, women who wish to become pregnant during the study period, women who cannot use birth control properly during the study period.
* Subject is considered as ineligible due to other factors by investigators.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
responder rate after deployment of valves | 6months after deployment of valves
  definition of responder: St. George's Respiratory Questionnaire (SGRQ) improving and Pulmonary Function improving (either Forced Expiratory Volume in 1 second (FEV1) improving or Inspiratory Capacity (IC) improving)

SECONDARY OUTCOMES:
Change in exercise capacity as measured by Six Minute Walk Test (6MWT) | before deployment of valves and 6months after deployment of valves
Change in dyspnea as measured by Baseline and Transition Dyspnea Indexes(BDI-TDI) | before deployment of valves and 6months after deployment of valves
Change in health status as measured by St. George's Respiratory Questionnaire(SGRQ) | before deployment of valves and 6months after deployment of valves
Change in dyspnea as measured by Medical Research Council, Modified (mMRC) Questionnaire | before deployment of valves and 6months after deployment of valves
Change in pulmonary function as measured by FEV1,Forced Vital Capacity(FVC),Vital Capacity(VC),Residual Volume(RV),IC,Total Lung Capacity(TLC),RV/TLC,Diffusing Capacity of the Lung for Carbon Monoxide(DLCO) | before deployment of valves and 6months after deployment of valves
Change in target lobe volume as measured by Quantitative CT (QCT) | before deployment of valves and 6months after deployment of valves

OTHER OUTCOMES:
Incidence of Severe and Serious Adverse Events(SAEs) whose relationship with the investigational device or the procedure cannot be ruled out | before deployment of valves and 6months after deployment of valves
Incidence of Adverse Events(AEs) whose relationship with the investigational device or the procedure cannot be ruled out | before deployment of valves and 6months after deployment of valves

CONTACTS AND LOCATIONS:
Locations (10):
- Japan (10):
  - Nagoya, Aichi-ken
  - Toyoake, Aichi-ken
  - Sapporo, Hokkaido
  - Kawasaki, Kanagawa
  - Matsusaka, Mie-ken
  - Mibu, Tochigi
  - Ube, Yamaguchi
  - Chiba
  - Fukuoka
  - Gifu